CLINICAL TRIAL: NCT04058639
Title: Diabetic Foot Ulcers: Shorter Treatment Period Using Custom Felt Relief?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/266
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Bandages; Wound Healing; Time; Relief
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- felt relief (Experimental): "custom felt relief"
  Interventions: Procedure: "custom felt relief"
- treatment as usual (Active Comparator): standard treatment usually provided by the Surgical Outpatient Clinic
  Interventions: Procedure: standard relief treatment

INTERVENTIONS:
Procedure: "custom felt relief" — Felt is adjusted to the wound by cutting it in different ways and layers once every week
  Arms: felt relief
Procedure: standard relief treatment — Felt in the shape of a letter U is put around the wound once every week.
  Arms: treatment as usual

SUMMARY:
The Surgical Outpatient Clinic at Molde Hospital has since 2015 offered specialized treatment for patients with diabetic foot ulcers. This treatment is given by an interdisciplinary diabetic foot ulcer team. The standard treatment for diabetic foot ulcers is relief, a method with good results.

Although the treatment as usual gives good results, the team wants to optimize this treatment. By using custom felt relief for each patient, the treatment period might be reduced considerably. The aim of this study is therefore to investigate whether custom felt relief gives shorter processing time compared to standard relief treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Diabetes Mellitus Type 1 or 2
* has neuropathic wounds under the foot
* understands and speaks Norwegian well
* competent to give consent

Exclusion Criteria:

* responds to the filament glue and/or the tape used in treatment
* in need of vascular surgery intervention
* to be admitted to the hospital
* in need of intravenously administered antibiotics due to wound infection.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
wound healing time in weeks | 2-8 weeks
  from the patients first visit (when the first felt dressing is applied) until the wound is healed

CONTACTS AND LOCATIONS:
Overall Officials: Tone Seim Fuglset, phd, Study Director — Helse Møre og Romsdal HF
Locations (1):
- Klinikk for Kirurgi Molde, Helse Møre og Romsdal HF, Molde, Norway

IPD SHARING:
Plan to Share IPD: No